CLINICAL TRIAL: NCT00485992
Title: Effectiveness of Utilizing Chlorhexidine Swabs for Accessing Lines and Results Impact on Catheter Related Blood Stream Infections in the Cardiac Intensive Care Unit
Brief Title: Chlorhexidine Swabs Effectiveness in Reducing Blood Stream Infections
Status: Terminated | Type: Observational
Why Stopped: sufficient data has been collected for significant conclusion
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Director Research, Children's Healthcare of Atlanta Institutional Review Board
Other Study IDs: 06-201
Record Dates: First submitted 2007-06-12; First posted 2007-06-13 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2008-01

CONDITIONS: Congenital Disorders
Keywords: blood stream infection; CICU; pediatric; chlorhexidine swabs
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Children's Healthcare of Atlanta (Children's) is collaborating with Child Health Corporation of America (CHCA) in the nationwide effort to reduce catheter related blood stream infections (BSIs). "As well as the human cost, central venous catheter related bloodstream infections significantly inflate hospital costs, mainly through increased length of stay in hospital, particularly in intensive care" (Jones, 2006).

The Cardiac Intensive Care Unit (CICU) is participating in this initiative by implementing the BSI "Bundles" per the CHCA guidelines. BSI "bundles" are a group of patient care practices designed to reduce BSI infection rates with implementation in patient care areas. The bundles include recommendations for central line maintenance including line insertion, dressing changes, line accesses, and monitoring for medical necessity. These bundles were implemented on January 16, 2006, when the BSI rate in the CICU had peaked at 18.2 (rate of infections per 1000 catheter days). The BSI rates historically for the past two years have been highly variable (see attached graph for data from Jan. 04 through Oct. 06). The target goal is to maintain a rate below 3.7 which has only been realized twice since the January BSI bundle implementation.

Current practice for the care of central lines outlined in the BSI Bundles is based on the Centers for Disease Control and Prevention (CDC) guidelines published in 2002. These guidelines included important changes to practice involving the use of chlorhexidine (CHG) containing products for improved infection prevention. CHG solutions are currently available as either 2% or 3.15% chlorhexidine gluconate in a 70% isopropyl alcohol solution.

The Primary Aim is to determine if CHG is effective as an antiseptic wipe for accessing lines to draw blood and administer medications. Compare the effectiveness of CHG containing alcohol wipes (3.15% CHG/70% isopropyl alcohol) to plain alcohol in order to determine best practice for the CICU.

DETAILED DESCRIPTION:
Children's Healthcare of Atlanta (Children's) is collaborating with Child Health Corporation of America (CHCA) in the nationwide effort to reduce catheter related blood stream infections (BSIs).

The Cardiac Intensive Care Unit (CICU) is participating in this initiative by implementing the BSI "Bundles" per the CHCA guidelines. BSI "bundles" are a group of patient care practices designed to reduce BSI infection rates with implementation in patient care areas.

Multiple risk factors are assumed to contribute to the high risk and rate of infection in the CICU patient population.

Many risk factors cannot be controlled, such as patient age, weight, diagnosis, etc. Hence the controllable risk factors are the focus for reducing BSI rates, primarily related to the care of central lines. This is the main focus of the BSI Bundles which are aimed at reducing the risks associated with the utilization of central lines.

The primary aim is to determine if CHG is effective as an antiseptic wipe for accessing lines to draw blood and administer medications. Compare the effectiveness of CHG containing alcohol wipes (3.15% CHG/70% isopropyl alcohol) to plain alcohol in order to determine best practice for the CICU.

The secondary aim is to reduce BSI rates in the CICU patient population, improving patient care outcomes and reducing costs of hospitalization by the resulting reduction and prevention of expected BSIs.

ELIGIBILITY:
Inclusion Criteria:

* Patients in Children's Healthcare of Atlanta, Egleston, in CICU between 8.1.06 to 12.31.06

Exclusion Criteria:

* those who do not qualify under inclusion criteria.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will observe from all children admitted to Children's CICU between 8.1.06 to 12.31.06; including both medical and surgical service patients.
Sampling Method: Non-Probability Sample
Enrollment: 352 (Actual)
Dates: Start 2006-08; Primary Completion 2006-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole M Jarrell, RNC, MSN, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States